CLINICAL TRIAL: NCT03073668
Title: The Effects of Pericardiotomy on Diastolic Reserve in Humans
Brief Title: Pericardial Resection to Treat Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Barry Borlaug, Associate Professor of Medicine, College of Medicine, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-000261
Record Dates: First submitted 2017-03-03; First posted 2017-03-08 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Heart Failure Patients (Experimental): After obtaining written informed consent, patients will undergo induction with general anesthesia as per clinical practice. The chest will be open but pericardium left intact. Cardiac hemodynamics will be measured using PA catheter already in place at rest, and then during conditions of increased cardiac preload, induced by passive leg elevation and saline bolus (300 ml administered over 1-2 minutes). The surgical team will perform anterior pericardiotomy. This will not be a complete pericardiectomy but rather a limited anterior incision to gain access to the heart for surgical exposure. The surgical team will then repeat hemodynamic assessments at rest and with acute volume loading (leg raise + saline) in exactly the same manner as with the pericardium intact.
  Interventions: Procedure: Anterior pericardiotomy; Drug: Saline

INTERVENTIONS:
Procedure: Anterior pericardiotomy — The surgical team will perform anterior pericardiotomy. This will not be a complete pericardiectomy but rather a limited anterior incision to gain access to the heart for surgical exposure.
Drug: Saline — During the measurement of cardiac hemodynamic tests, a saline bolus of 300 ml will be administered over 1-2 minutes.

SUMMARY:
The researchers are doing this study to find out whether there will be less increase in cardiac filling pressure after the surgeon opens the pericardium (the membrane around the heart) than when the pericardium is intact. The researchers want to see whether opening the pericardium is an effective way to reduce the blood filling pressures in the heart.

DETAILED DESCRIPTION:
This study will enroll patients with risk factors for LV diastolic dysfunction, either coronary artery disease or aortic stenosis, who are already undergoing cardiac surgery for clinical purposes (e.g. coronary artery bypass grafting or valvular heart disease).

Hemodynamic tests will be performed using standard clinical resources used as part of routine care in this setting, including pulmonary artery (PA) catheterization. After obtaining written informed consent, patients will undergo induction with general anesthesia as per clinical practice. The chest will be open but pericardium left intact. Cardiac hemodynamics (PA wedge pressure, PAWP; PA pressure, PAP, right atrial pressure, RAP) will be measured using PA catheter already in place at rest, and then during conditions of increased cardiac preload, induced by passive leg elevation and saline bolus (300 ml administered over 1-2 minutes).

The surgical team will then perform anterior pericardiotomy, with removal of pericardial restraint similar to our percutaneous approach but using currently-available surgical tools. This will not be a complete pericardiectomy but rather a limited anterior incision to gain access to the heart for surgical exposure (standard care).

The surgical team will then repeat hemodynamic assessments at rest and with acute volume loading (leg raise + saline) in exactly the same manner as with the pericardium intact. Our hypothesis is that as compared to pericardium intact, the increase in PAWP with volume loading will be reduced following opening of the pericardium.

ELIGIBILITY:
Inclusion

* >17 years old
* Subjects having open sternotomy for either aortic valve stenosis or coronary artery bypass grafting (or both)
* Provide informed consent Exclusion
* <18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2018-01-23 (Actual); Study Completion 2019-02-02 (Actual)

PRIMARY OUTCOMES:
Change in Pulmonary Artery Wedge Pressure (PAWP) | Baseline, approximately 1 hour
  Patients will undergo induction with general anesthesia, and at baseline the chest will be open, but pericardium left intact. Cardiac hemodynamics will be measured using the Pulmonary Artery Catheter already in place. The surgical team will then perform anterior pericardiotomy, with removal of pericardial restraint, and cardiac hemodynamics will be measured again.

SECONDARY OUTCOMES:
Change in Pulmonary Artery Pressure (PAP) | Baseline, approximately 1 hour
  Patients will undergo induction with general anesthesia, and at baseline the chest will be open, but pericardium left intact. Cardiac hemodynamics will be measured using the Pulmonary Artery Catheter already in place. The surgical team will then perform anterior pericardiotomy, with removal of pericardial restraint, and cardiac hemodynamics will be measured again.
Change in Right Arterial Pressure (RAP) | Baseline, approximately 1 hour
  Patients will undergo induction with general anesthesia, and at baseline the chest will be open, but pericardium left intact. Cardiac hemodynamics will be measured using the Pulmonary Artery Catheter already in place. The surgical team will then perform anterior pericardiotomy, with removal of pericardial restraint, and cardiac hemodynamics will be measured again.

CONTACTS AND LOCATIONS:
Overall Officials: Barry A Borlaug, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials